CLINICAL TRIAL: NCT04211389
Title: A Phase 3, 8-Week, Parallel Group, Double Blind, Vehicle-Controlled Study of the Safety and Efficacy of ARQ-151 Cream 0.3% Administered QD in Subjects With Chronic Plaque Psoriasis
Brief Title: Twin Trial of PDE4 Inhibition With Roflumilast for the Management of Plaque Psoriasis
Acronym: DERMIS-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARQ-151-302
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Results first posted 2022-10-18 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Chronic Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARQ-151 cream 0.3% (Active Comparator): Active comparator
  Interventions: Drug: ARQ-151 0.3% cream
- ARQ-151 cream vehicle (Placebo Comparator): Placebo comparator
  Interventions: Drug: ARQ-151 vehicle cream

INTERVENTIONS:
Drug: ARQ-151 0.3% cream — ARQ-151 0.3% cream
  Arms: ARQ-151 cream 0.3%
Drug: ARQ-151 vehicle cream — ARQ-151 vehicle cream
  Arms: ARQ-151 cream vehicle

SUMMARY:
This study will assess the safety and efficacy of ARQ-151 cream vs placebo applied once a day for 56 days by subjects with chronic plaque psoriasis

DETAILED DESCRIPTION:
This is a parallel group, double blind, vehicle-controlled study in which ARQ-151 cream or vehicle is applied once daily x 8 weeks to subjects with psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Participants legally competent to sign and give informed consented and if appropriate assent as required by local laws
* Males and females ages 2 years and older (inclusive)
* Clinical diagnosis of psoriasis vulgaris of at least 6 months duration (3 months for children) as determined by the Investigator
* Females of childbearing potential (FOCBP) must have a negative pregnancy test at Screening (Visit 1) and Baseline (Visit 2). In addition, sexually active FOCBP must agree to use at least one form of highly effective contraception throughout the trial.
* In good health as judged by the Investigator, based on medical history, physical examination, serum chemistry labs, hematology values, and urinalysis.
* Subjects considered reliable and capable of adhering to the Protocol and visit schedule, according to the judgment of the Investigator.

Exclusion Criteria:

* Planned excessive exposure of treated area(s) to either natural or artificial sunlight, tanning bed or other LED.

  * Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.
  * Previous treatment with ARQ-151 or its active ingredient
  * Subjects with any serious medical condition or laboratory abnormality that would prevent study participation or place the subject at significant risk, as determined by the Investigator.
  * Subjects with a history of chronic alcohol or drug abuse within 6 months of initiation of investigational product
  * Subjects who are unable to communicate, read or understand the local language, or who display another condition, which in the Investigator's opinion, makes them unsuitable for clinical study participation

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (39):
- United States (31):
  - Arcutis Biotherapeutics Clinical Site 203, Scottsdale, Arizona
  - Arcutis Biotherapeutics Clinical Site 239, Beverly Hills, California
  - Arcutis Biotherapeutics Clinical Site 225, Encino, California
  - Arcutis Biotherapeutics Clinical Site 220, San Diego, California
  - Arcutis Biotherapeutics Clinical Site 208, Santa Monica, California
  - Arcutis Biotherapeutics Clinical Site 215, Santa Monica, California
  - Arcutis Biotherapeutics Clinical Site 223, Boynton Beach, Florida
  - Arcutis Biotherapeutics Clinical Site 237, DeLand, Florida
  - Arcutis Biotherapeutics Clinical Site 228, Largo, Florida
  - Arcutis Biotherapeutics Clinical Site 201, North Miami Beach, Florida
  - Arcutis Biotherapeutics Clinical Site 209, Sweetwater, Florida
  - Arcutis Biotherapeutics Clinical Site 214, Indianapolis, Indiana
  - Arcutis Biotherapeutics Clinical Site 217, Louisville, Kentucky
  - Arcutis Biotherapeutics Clinical Site 211, Lake Charles, Louisiana
  - Arcutis Biotherapeutics Clinical Site 213, Metairie, Louisiana
  - Arcutis Biotherapeutics Clinical Site 224, New Orleans, Louisiana
  - Arcutis Biotherapeutics Clinical Site 212, Detroit, Michigan
  - Arcutis Biotherapeutics Clinical Site 216, Fridley, Minnesota
  - Arcutis Biotherapeutics Clinical Site 227, Saint Joseph, Missouri
  - Arcutis Biotherapeutics Clinical Site 219, Las Vegas, Nevada
  - Arcutis Biotherapeutics Clinical Site 231, Las Vegas, Nevada
  - Arcutis Biotherapeutics Clinical Site 240, Reno, Nevada
  - Arcutis Biotherapeutics Clinical Site 236, Portsmouth, New Hampshire
  - Arcutis Biotherapeutics Clinical Site 222, Oklahoma City, Oklahoma
  - Arcutis Biotherapeutics Clinical Site 229, Broomall, Pennsylvania
  - Arcutis Biotherapeutics Clinical Site 233, Knoxville, Tennessee
  - Arcutis Biotherapeutics Clinical Site 221, Murfreesboro, Tennessee
  - Arcutis Biotherapeutics Clinical Site 206, Arlington, Texas
  - Arcutis Biotherapeutics Clinical Site 238, Houston, Texas
  - Arcutis Biotherapeutics Clinical Site 210, West Jordan, Utah
  - Arcutis Biotherapeutics Clinical Site 230, Richmond, Virginia
- Canada (8):
  - Arcutis Biotherapeutics Clinical Site 207, Surrey, British Columbia
  - Arcutis Biotherapeutics Clinical Site 226, Surrey, British Columbia
  - Arcutis Biotherapeutics Clinical Site 232, Winnepeg, Manitoba
  - Arcutis Biotherapeutics Clinical Site 234, Fredericton, New Brunswick
  - Arcutis Biotherapeutics Clinical Site 205, Ajax, Ontario
  - Arcutis Biotherapeutics Clinical Site 218, Barrie, Ontario
  - Arcutis Biotherapeutics Clinical Site 235, Toronto, Ontario
  - Arcutis Biotherapeutics Clinical Site 204, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Papp KA, Del Rosso JQ, Lebwohl MG, Gooderham MJ, Hebert AA, Hong HC, Kircik LH, Pariser DM, Stein Gold L, Strober B, Seal MS, Krupa D, Chu DH, Burnett P, Berk DR, Higham RC. Roflumilast Cream 0.3% in Patients with Chronic Plaque Psoriasis: Pooled PASI and PASI-HD Results from the DERMIS Phase III Trials. Dermatol Ther (Heidelb). 2025 Dec;15(12):3733-3744. doi: 10.1007/s13555-025-01562-4. Epub 2025 Oct 24. PMID 41134450
- [Derived] Thurston AW Jr, Osborne DW, Snyder S, Higham RC, Burnett P, Berk DR. Pharmacokinetics of Roflumilast Cream in Chronic Plaque Psoriasis: Data from Phase I to Phase III Studies. Am J Clin Dermatol. 2023 Mar;24(2):315-324. doi: 10.1007/s40257-022-00741-9. Epub 2022 Nov 24. PMID 36422852
- [Derived] Lebwohl MG, Kircik LH, Moore AY, Stein Gold L, Draelos ZD, Gooderham MJ, Papp KA, Bagel J, Bhatia N, Del Rosso JQ, Ferris LK, Green LJ, Hebert AA, Jones T, Kempers SE, Pariser DM, Yamauchi PS, Zirwas M, Albrecht L, Devani AR, Lomaga M, Feng A, Snyder S, Burnett P, Higham RC, Berk DR. Effect of Roflumilast Cream vs Vehicle Cream on Chronic Plaque Psoriasis: The DERMIS-1 and DERMIS-2 Randomized Clinical Trials. JAMA. 2022 Sep 20;328(11):1073-1084. doi: 10.1001/jama.2022.15632. PMID 36125472

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult participants with chronic plaque psoriasis were enrolled at 43 study sites in the United States and Canada.
Groups:
- Roflumilast Cream 0.3%: Participants applied roflumilast cream 0.3% QD for 8 weeks. There was a 1-week follow-up period after completing treatment.
- Vehicle Cream: Participants applied inactive vehicle cream matched to roflumilast cream QD for 8 weeks. There was a 1-week follow-up period after completing treatment.
Period: Overall Study
Arm/Group | Roflumilast Cream 0.3% | Vehicle Cream
Started | 290 | 152
Completed | 264 | 131
Not Completed | 26 | 21
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 15 | 7
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast Cream 0.3% | Vehicle Cream | Total
Number analyzed (Participants) | 290 | 152 | 442
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (15.07) | 47.1 (14.07) | 47.0 (14.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 52 | 166
  Male | 176 | 100 | 276
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 76 | 50 | 126
  Not Hispanic or Latino | 213 | 102 | 315
  Unknown or Not Reported | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American-Indian or Alaska Native | 0 | 1 | 1
  Asian | 20 | 9 | 29
  Black or African American | 13 | 9 | 22
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  White | 240 | 126 | 366
  Not Reported | 5 | 2 | 7
  Other | 8 | 4 | 12
  More than 1 Race | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 76 | 50 | 126
  Not Hispanic or Latino | 213 | 102 | 315
  Not Reported | 1 | 0 | 1
Investigator Global Assessment (IGA) Scores at Baseline [Count of Participants; unit: Participants] — The IGA is 5-point scale assessing the severity of plaque psoriasis, with scores ranging from 0 ('clear') to 4 ('severe'), with higher scores indicating greater plaque severity.
  Participants
    0 - Clear | 0 | 0 | 0
    1 - Almost Clear | 0 | 0 | 0
    2 - Mild | 50 | 24 | 74
    3 - Moderate | 220 | 118 | 338
    4 - Severe | 20 | 10 | 30
Psoriasis Area Severity Index (PASI) Score [Mean (Standard Deviation); unit: score on a scale] — The Psoriasis Area and Severity Index (PASI) is widely used for the measurement of severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range from 0 (no disease) to 72 (maximal disease), with higher scores indicating greater symptom severity
  score on a scale | 6.5 (3.22) | 7.0 (3.52) | 6.7 (3.33)
Worst Itch Numerical Rating Scale (WI-NRS) Baseline Score [Mean (Standard Deviation); unit: units on a scale] — The WI-NRS is a simple, single item scale to assess the participant-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the participant experienced in the past 24 hours. Higher scores indicate greater symptom severity.
  units on a scale | 5.8 (2.61) | 6.1 (2.75) | 5.9 (2.66)
Baseline Psoriasis Symptom Diary (PSD) Total Score [Mean (Standard Deviation); unit: score on a scale] — The PSD is a 16-item questionnaire asking subjects to rate the severity of psoriasis-related symptoms in the past 24 hours. Each question is scored from 0 ("no symptoms") to 10 ("worst imaginable symptoms"). Scores range from 0 to 160, with higher scores indicating greater symptom severity.
  score on a scale | 69.3 (40.66) | 77.4 (41.24) | 72.1 (41.00)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Success on the Investigator Global Assessment (IGA) Scale
Description: The number of participants achieving "success" in IGA assessment of disease severity at Week 8 is presented for each arm. Success was defined as achievement of an IGA score of 0 ('clear') or 1 ('almost clear') at Week 8, accompanied by a ≥2-grade improvement from baseline IGA score. The IGA is 5-point scale assessing the severity of plaque psoriasis, with scores ranging from 0 ('clear') to 4 ('severe'), and higher scores indicate greater symptom severity. The IGA scores are based on observed data, whereas odds ratio and p-values were calculated using multiple imputation of missing values.
Time Frame: Week 8
Population: All randomized participants with data are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Cream 0.3% | Vehicle Cream
Number analyzed (Participants) | 264 | 131
Participants | 99 | 9
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; IGA Success at Week 8 Odds Ratio; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Stratification by pooled study site, baseline IGA, and baseline intertriginous involvement per randomization with multiple imputation of missing data; Odds Ratio (OR) = 6.59, 95% CI 2-sided [3.17 to 13.70] — Common OR stratified by pooled study site, baseline IGA, and baseline intertriginous involvement per randomization with multiple imputation of missing data

2. Secondary Outcome: Time to Achieve Psoriasis Area Severity Index-50 (PASI-50)
Description: The Psoriasis Area and Severity Index (PASI) is widely used for the measurement of severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range from 0 (no disease) to 72 (maximal disease), with higher scores indicating greater symptom severity. The time to achieve PASI-50 (defined as a 50% reduction from baseline in PASI score) is presented, and is based on observed data only. Participants are included whether they achieved PASI-50 or not.
Time Frame: From start of treatment to achievement of PASI-50 or study completion/early termination (maximum duration = 124 days)
Population: All randomized participants are included.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Roflumilast Cream 0.3% | Vehicle Cream
Number analyzed (Participants) | 290 | 152
days | 30.0 [29.0 to 42.0] | NA [71.0 to NA] — Median number of days and upper bound of CI were not calculable due to low number of cases.
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Time to Achieve PASI-50; Test type: Superiority; p < 0.0001, Log Rank; Unstratified log-rank test; Hazard Ratio (HR) = 4.207, 95% CI 2-sided [3.029 to 5.844] — HR stratified by pooled study site, baseline IGA, and baseline intertriginous involvement per randomization

3. Secondary Outcome: Number of Participants Achieving Psoriasis Area Severity Index-75 (PASI-75)
Description: The Psoriasis Area and Severity Index (PASI) is widely used for the measurement of severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range from 0 (no disease) to 72 (maximal disease), with higher scores indicating greater symptom severity. The number of participants achieving PASI-75 (defined as a 75% reduction from baseline in PASI score) at Week 8 is presented. Participant counts are based on observed data only.
Time Frame: Baseline (Day 1) and Week 8
Population: All randomized participants with data available are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Cream 0.3% | Vehicle Cream
Number analyzed (Participants) | 264 | 131
Participants | 103 | 7
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; PASI-75 at Week 8 Odds Ratio; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study site, baseline IGA, and baseline intertriginous involvement per randomization with multiple imputation of missing data; Odds Ratio (OR) = 10.42, 95% CI 2-sided [4.49 to 24.19] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants Achieving Psoriasis Area Severity Index-90 (PASI-90)
Description: The Psoriasis Area and Severity Index (PASI) is widely used for the measurement of severity of psoriasis. PASI combines the assessment of the severity of lesions and the area affected into a single score in the range from 0 (no disease) to 72 (maximal disease), with higher scores indicating greater symptom severity. The number of participants achieving PASI-90 (defined as a 90% reduction from baseline in PASI score) at Week 8 is presented. Participant counts are based on observed data only.
Time Frame: Baseline (Day 1) and Week 8
Population: All randomized participants with data available are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Cream 0.3% | Vehicle Cream
Number analyzed (Participants) | 290 | 152
Participants | 45 | 3
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; PASI-90 at Week 8 Odds Ratio; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 8.51, 95% CI 2-sided [2.45 to 28.86] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants Achieving Success in Intertriginous Investigator Global Assessment (I-IGA) Scale Assessment of Disease Severity at Week 8
Description: The number of participants with I-IGA score ≥2 at baseline achieving "success" in IGA assessment of disease severity at Week 8 is presented (observed data only) for each arm. Success was defined as achievement of an I-IGA score of 0 ('clear') or 1 ('almost clear') at Week 8, accompanied by a ≥2-grade improvement from baseline I-IGA score. The IGA is a 5-point scale assessing the severity of plaque psoriasis, with scores ranging from 0 ('clear') to 4 ('severe'), and higher scores indicate greater symptom severity.
Time Frame: Week 8
Population: All randomized participants with intertriginous area involvement and I-IGA score at Baseline ≥ 2 who have Week 8 data available are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Cream 0.3% | Vehicle Cream
Number analyzed (Participants) | 47 | 27
Participants | 32 | 5
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; I-IGA Success at Week 8 Odds Ratio; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel; Stratified by pooled study site and baseline IGA per randomization with multiple imputation of missing data; Odds Ratio (OR) = 11.18, 95% CI 2-sided [2.33 to 53.68] — Common OR stratified by pooled study site and baseline IGA per randomization with multiple imputation of missing data

6. Secondary Outcome: Number of Participants Achieving I-IGA Score of 'Clear' at Week 8
Description: The number of participants achieving an IGA score of 0 ('clear') at Week 8 is presented (observed data only) for each arm. The I-IGA is a 5-point scale assessing the severity of intertriginous area plaque psoriasis, with scores ranging from 0 ('clear') to 4 ('severe'), and higher scores indicate greater symptom severity.
Time Frame: Week 8
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Cream 0.3% | Vehicle Cream
Number analyzed (Participants) | 47 | 27
Participants | 27 | 2
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; I-IGA Clear at Week 8 Odds Ratio; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Stratified by pooled study site and baseline IGA with multiple imputation of missing data; Odds Ratio (OR) = 15.27, 95% CI 2-sided [3.10 to 75.35] — Common odds ratio stratified by pooled study site and baseline IGA with multiple imputation of missing data

7. Secondary Outcome: Number of Participants Achieving Success in Worst Itch Numerical Rating Scale (WI-NRS) Pruritus Score
Description: The number of participants achieving success in WI-NRS is presented. Success is defined as achievement of a ≥ 4-point reduction in WI-NRS pruritus score in participants with WI-NRS pruritus score ≥ 4 at baseline. The WI-NRS is a 10 point scale ranging from 0 ('no itch') to 10 ('worst itch imaginable') the participant experienced in the past 24 hours, with higher scores indicating greater symptoms severity. Results are based on observed data only.
Time Frame: Baseline (Day 1) and Week 2, Week 4, Week 8
Population: All randomized participants with WI-NRS pruritus score ≥4 at baseline and data available at the relevant time points are included.
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Cream 0.3% | Vehicle Cream
Number analyzed (Participants) | 215 | 109
Participants
  Week 2 | 90 | 23
  Week 4: number analyzed (Participants) | 212 | 105
  Week 4 | 120 | 23
  Week 8: number analyzed (Participants) | 206 | 101
  Week 8 | 143 | 36
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Test type: Superiority — WI-NRS Success at Week 2 Odds Ratio; p = 0.0026, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 2.56, 95% CI 2-sided [1.43 to 4.58] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Test type: Superiority — WI-NRS Success at Week 4 Odds Ratio; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 4.93, 95% CI 2-sided [2.65 to 9.18] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; Test type: Superiority — WI-NRS Success at Week 8 Odds Ratio; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 3.59, 95% CI 2-sided [2.07 to 6.23] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline in Psoriasis Symptoms Diary (PSD) Score
Description: The PSD is a 16-item questionnaire asking subjects to rate the severity of psoriasis-related symptoms in the past 24 hours. Each question is scored from 0 ("no symptoms") to 10 ("worst imaginable symptoms"). Scores range from 0 to 160, with higher scores indicating greater symptom severity. The least squares (LS) mean (95% CI) change in PSD total score relative to baseline is presented for each treatment arm, with decreases from baseline indicating symptom improvement.
Time Frame: Baseline (Day 1) and Weeks 4 and 8
Population: All randomized participants are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Roflumilast Cream 0.3% | Vehicle Cream
Number analyzed (Participants) | 290 | 152
score on a scale
  Week 4: number analyzed (Participants) | 262 | 135
  Week 4 | -42.7 [-47.7 to -37.7] | -16.7 [-22.8 to -10.6]
  Week 8: number analyzed (Participants) | 257 | 127
  Week 8 | -49.3 [-54.8 to -43.7] | -22.8 [-29.6 to -16.0]
Statistical Analysis 1: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; LS Mean Difference at Week 4; Test type: Superiority; p < 0.0001, ANCOVA; Site, baseline IGA, baseline intertriginous involvement, and baseline PSD scores were independent variables, multiple imputation used for missing data; Mean Difference (Final Values) = -26.0, 95% CI 2-sided [-31.9 to -20.0] — Site, baseline IGA, baseline intertriginous involvement, and baseline PSD scores were independent variables, multiple imputation used for missing data
Statistical Analysis 2: Comparison: Roflumilast Cream 0.3% vs Vehicle Cream; LS Mean Difference at Week 8; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -26.5, 95% CI 2-sided [-33.2 to -19.7] — [estimate comment as in outcome 8, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to 124 days
Description: All participants who received ≥1 dose of study treatment are included.
Arm/Group | Roflumilast Cream 0.3% | Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/290 | 0/152
Serious Adverse Events (participants affected / at risk) | 0/290 | 1/152
Other Adverse Events (participants affected / at risk) | 0/290 | 0/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Roflumilast Cream 0.3% (N=290) | Vehicle Cream (N=152)
Cervical radiculopathy (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor is supportive of publishing clinical trial findings. The process of coordinating publication efforts is detailed in the Clinical Trial Agreement.

DOCUMENTS (2):
  • Study Protocol (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/89/NCT04211389/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT04211389/SAP_001.pdf